CLINICAL TRIAL: NCT03962660
Title: Randomized Controlled Trial of Harm Reduction for Tobacco Smoking With Support of Tobacco-Replacing Electronic Nicotine Delivery Systems (HaRTS-TRENDS)
Brief Title: Harm Reduction for Tobacco Smoking With Support of Tobacco-Replacing Electronic Nicotine Delivery Systems
Acronym: HaRTS-TRENDS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Washington (Other)
Collaborators: Downtown Emergency Service Center (Unknown); Washington State University (Other)
Responsible Party: Principal Investigator, Susan Collins, Associate Professor, School of Medicine: Psychiatry, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00006430
Record Dates: First submitted 2019-05-17; First posted 2019-05-24 (Actual); Last update posted 2019-05-24 (Actual); Status verified 2019-05

CONDITIONS: Smoking, Tobacco
MeSH Terms: conditions — Tobacco Smoking | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: HaRTS-TRENDS, in which participants will attend 4, 30-minute sessions with research staff. They will discuss participants' current smoking and their goals around reducing smoking-related harm and improving their health-related quality of life. Participants will also engage in discussions about the safety profiles of different nicotine products. One group of these products, e-cigarettes, is 95% safer than smoking and will be made available to participants to help them achieve their harm-reduction goals. They will receive instructions and demonstrations for its safe and proper use.
  -OR-
  Standard care, in which will attend 4, 30-minute sessions of brief advice to quit.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HaRTS-TRENDS (Experimental): See description below.
  Interventions: Other: HaRTS-TRENDS
- Standard Care (SC) (Active Comparator): See description below.
  Interventions: Other: Standard Care (SC)

INTERVENTIONS:
Other: HaRTS-TRENDS — HaRTS-TRENDS comprises 4, individual sessions delivered in the context of the interventionist's pragmatic harm-reduction mindset paired with a compassionate, advocacy-oriented "heart-set" or style. It comprises the delivery of 4 manualized components, including a) participant-led tracking of preferred smoking outcomes, b) elicitation of participants' harm-reduction goals and their progress toward achieving them, c) discussion of the relative risks of various nicotine delivery systems, and d) instruction in using ENDS. Additionally, HaRTS-TRENDS entails provision of commercially available ENDS.
  Arms: HaRTS-TRENDS
Other: Standard Care (SC) — The 4-session, individual standard care control condition entails the well-documented and evidence-based 5 As intervention (i.e., Ask about nicotine use, Assess use, Advise to quit smoking, Assist with exploring current smoking/planning smoking cessation, Arrange follow-up). Part of arranging follow-up is the recommendation to call the smoking quit line, which can supply additional counseling and nicotine replacement therapy.
  Other Names: 5 As
  Arms: Standard Care (SC)

SUMMARY:
This study will evaluate the effectiveness of HaRTS-TRENDS compared to standard care (i.e., brief advice to quit + referral to state quit line that offers free NRT) in facilitating a biochemically verified nonsmoking and b) reducing smoking-related harm as measured by concentration of urinary tobacco-specific nitrosamines (TSNAs). Potential underlying mechanisms of changes in the proposed outcomes--including nicotine craving and smoking reduction, respectively--will be tested.

DETAILED DESCRIPTION:
The prevalence of smoking and smoking-related illness is disproportionately higher among people experiencing chronic homelessness than among people in the general population. Unfortunately, smoking cessation treatment does not reach or engage the overwhelming majority of smokers experiencing chronic homelessness, and smoking-related harm persists even after people are housed. There have therefore been calls for more flexible and client-centered approaches tailored to this population's needs. In response, we are proposing a randomized controlled trial (RCT) of Harm-Reduction for Tobacco Smoking with support of Tobacco-Replacing Electronic Nicotine Delivery Systems (HaRTS-TRENDS) as an innovative, empirically informed, and client-driven alternative to traditional smoking cessation treatment. To maximize its efficacy, the 4-session, individual HaRTS-TRENDS was collaboratively designed with a community advisory board made up of researchers, people with lived experience of chronic homelessness and smoking, and staff and management at a nonprofit, community-based housing agency. HaRTS-TRENDS entails the provision of electronic nicotine delivery systems (ENDS) in conjunction with harm-reduction counseling. Interventionists embody a compassionate, advocacy-oriented "heart-set" or style and deliver manualized components that include a) participant-led tracking of preferred smoking outcomes, b) elicitation of participants' harm-reduction goals and their progress toward achieving them, c) discussion of the relative risks of various nicotine delivery systems, and d) instruction in using ENDS. The proposed study will feature a randomized controlled trial (N=94) of HaRTS-TRENDS among smokers with lived experience of chronic homelessness who have moved into permanent, supportive housing. Participants will be randomized to receive HaRTS-TRENDS or standard care. The standard care, which is what people most commonly receive from providers, is brief advice to quit plus referral to the Washington State quitline where participants have access to free NRT. All participants will be assessed at baseline and posttest as well as at 1-, 3-, 6-, and 12-month follow-ups. Analyses will be conducted to test the efficacy of HaRTS-TRENDS compared to SC in a) facilitating biochemically verified nonsmoking and b) reducing smoking-related harm as measured by concentration of urinary tobacco-specific nitrosamines (TSNAs). It is hypothesized that, compared to SC participants, HaRTS-TRENDS participants will show a significantly greater likelihood of nonsmoking and reduced concentration of TSNAs. Further, we will examine reductions in smoking craving as a mediator of the HaRTS-TRENDS effect on nonsmoking as well as nonsmoking as a mediator of the HaRTS-TRENDS effect on TSNA concentration. If its results are positive, this project will lay the groundwork for longer-term objectives including dissemination of HaRTS-TRENDS to researchers, clinicians, and community-based agencies to decrease smoking-related harm for a high-cost and severely affected population.

ELIGIBILITY:
Inclusion Criteria:

* Having a history of chronic homelessness according to the widely accepted federal definition,
* Being a current DESC client living in one of DESC's participating permanent supportive housing projects,
* Being between 21-65 years of age,
* Being a daily smoker (>4 cigarettes/day in the past year with a breath CO ≥ 6 ppm or salivary cotinine test at level 1 if CO < 6 ppm)
* Having adequate English language skills to understand verbal information and communicate in the study

Exclusion Criteria:

* Use of other tobacco products besides cigarettes ≥ 9 days in the past month
* Refusal or inability to consent to participation in research
* Constituting a risk to the safety and security of other clients or staff.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2019-05-09 (Actual); Primary Completion 2021-04-30 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Nonsmoking | Change across the 12-month follow-up
  Biologically verified nonsmoking (i.e., self-reported nonsmoking if corresponding CO measure is < 8) in the past 7 days will serve as a primary outcome as well as a potential mediator of the HaRTS-TRENDS effect on TSNA concentration.
TSNA Concentration | Change across the 12-month follow-up
  This primary outcome entails urinary concentration of a tobacco-specific nitrosamine (i.e., NNK), a key carcinogen in tobacco. Secondarily, TSNA concentration will be used as a longer-term biochemical index of tobacco use.

SECONDARY OUTCOMES:
smoking intensity | Change across the 12-month follow-up
  Self-reported smoking intensity is the mean number of cigarettes participants report smoking per day in the 7 days prior to the assessment.
smoking frequency | Change across the 12-month follow-up
  Self-reported smoking frequency is the number of days participants report smoking in the 7 days prior to the assessment.
CO level | Change across the 12-month follow-up
  Carbon monoxide in exhaled air will be examined secondarily as a continuous measure of reduced smoking-related harm. It will also be used to biochemically verify the 7-day nonsmoking primary outcome.
cotinine levels | Change across the 12-month follow-up
  Urinary cotinine will reflect participants' recent nicotine use.
FEV1% | Change across the 12-month follow-up
  FEV1% is the ratio of predicted lung capacity based on participants' height, age and gender with participants' forced expiratory volume in the first second of expiration as a percentage of the predicted value.
Clinical COPD questionnaire | Change across the 12-month follow-up
  The 10-item Clinical COPD Questionnaire will be used to calculate an overall summary score representing respiratory HR-QoL over 3 domains: respiratory symptoms (e.g., shortness of breath), functional state (e.g., ability to climb stairs), and mental state (i.e., concern about getting a cold or breathing getting worse). The total score is calculated by summing the scores of the individual items and dividing by 10 (the number of individual items) giving a total score between 0 and 6 with higher scores representing worse HRQoL.
EQ-5D-5L | Change across the 12-month follow-up
  This self-report measure yields 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Additionally, the EuroQoL-Visual Analog Scale (EQ-VAS) is a single item representing health-related quality of life via participants' general assessments of their current health, where 0 = the worst health imaginable and 100 = the best health imaginable.

OTHER OUTCOMES:
smoking craving | Change across the 12-month follow-up
  Smoking craving is a potential mediator of the proposed intervention effects and will be measured using the Questionnaire for Smoking Urges-Brief (QSU-B) consists of 10 items rated on 7-point Likert scales ranging from 0 (strongly disagree) to 6 (strongly agree). Changes in smoking craving summary scores will be tested as a mediator of the HaRTS-TRENDS effects on complete switchover.
side effects of ENDS | Change across the 12-month follow-up
  We will assess participants' experience of known, ENDS-related adverse events (i.e., dry mouth, throat irritation, short-ness of breath, headache, cough, tachycardia, nausea) using a 5-item, 5-point Likert-type questionnaire (ranging from 0=none to 5=severe) that was adapted from the Systematic Assessment for Treatment Emergent Effects (SAFTEE) interview.

CONTACTS AND LOCATIONS:
Overall Officials: Susan E Collins, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Washington - Harborview Medical Center, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No
The proposed research will involve people recruited from prominent Housing First programs serving chronically homeless people who are often multiply affected by psychiatric, medical and substance-use disorders. The proposed sample will be recruited from a highly vulnerable and marginalized population in a tight-knit urban community. Furthermore, the partnering agency is well-known for its housing approach, and regularly conducts tours to help inform other housing providers, policy makers, and other public stakeholders about this model to promote replicability. Thus, even with the removal of all identifiers, we believe that it could become difficult to fully protect the identities of participants and their data (including e-cigarette use and smoking which are not currently allowed in housing). For these reasons, we do not have immediate plans to share the data collected in the context of the proposed study.